CLINICAL TRIAL: NCT02768194
Title: Assessment of Dentine Tubule Occlusion in a Modified in Situ Model
Brief Title: Dentine Tubule Occlusion Assessment in a Modified in Situ Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 205699
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-03

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — fluorophosphate; Mineral Waters

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Test Product (0.454% stannous fluoride) (Experimental): Participants will use dentifrice containing 0.454% stannous fluoride. Appliances brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily will be then returned to the participant's mouth. Each appliance will be brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances will be returned to the participant's mouth and the participant will rinse with 10 mls of mineral water for 5 seconds.
  Interventions: Device: Stannous fluoride
- Reference Product (0.76% sodium monofluorophosphate) (Active Comparator): Participants will use dentifrice containing 0.76% sodium monofluorophosphate. Appliances brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily will be then returned to the participant's mouth. Each appliance will be brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances will be returned to the participant's mouth and the participant will rinse with 10 mls of mineral water for 5 seconds.
  Interventions: Other: Sodium monofluorophosphate
- Negative Control (Mineral water) (Other): Participants will use commercially available mineral water. Appliances brushed ex situ in mineral water twice daily will be then returned to the participant's mouth. Each appliance will be brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in mineral water. Appliances will be returned to the participant's mouth and the participant will rinse with 10 mls of mineral water for 5 seconds.
  Interventions: Other: Mineral water

INTERVENTIONS:
Device: Stannous fluoride — Dentifrice containing 0.454% stannous fluoride
  Arms: Test Product (0.454% stannous fluoride)
Other: Sodium monofluorophosphate — Dentifrice containing 0.76% sodium monofluorophosphate
  Arms: Reference Product (0.76% sodium monofluorophosphate)
Other: Mineral water — Commercially available mineral water
  Arms: Negative Control (Mineral water)

SUMMARY:
This will be a single centre, single blind, randomized, three treatment, three period crossover design, modified, in situ, study in healthy participants. In this in situ model the tubule occlusion properties of dentifrices will be evaluated by comparing an experimental dentifrice formulation to a regular fluoride dentifrice and a negative control (mineral water) over a ten day period.

DETAILED DESCRIPTION:
This modified in situ model study will evaluate the mode-of-action of an experimental dentifrice containing stannous fluoride to occlude tubules compared to a regular fluoride dentifrice and a negative control (mineral water). The study treatments will be administered for a total of 10 days, with participants wearing two appliances in their mouth that will hold samples of dentine. The dentine samples will be examined after 1, 4, 8 and 10 days of treatment using scanning electron microscopy (SEM) and the resulting images graded for the amount of occlusion. In addition, the robustness of any occlusion generated by the treatments will be tested by exposing the dentine samples to an acid challenge (orange juice) after 9 and 10 days treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 and 80 years
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination, absence of any condition that would impact on the participant's safety or well being or affect the individual's ability to understand and follow procedures and requirements.
* Be able to accommodate the lower bi-lateral buccal intra-oral appliances each fitted with four dentine samples

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding
* Current or recurrent disease/dental pathology that in the opinion of the investigator could affect the study outcomes.

Current susceptibility to acid regurgitation, any orthodontic appliances, restorations, bridgework or dentures that in the opinion of the investigator would interfere with the study outcomes, recurrent or regular aphthous ulcers, severe gingivitis, carious lesions and periodontal disease,signs of severe dental erosion, any condition or medication which in the opinion of the investigator is currently causing xerostomia, and individuals who require antibiotic prophylaxis for dental procedures

* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another study (clinical or cosmetic studies) or receipt of an investigational drug within 15 days of the screening visit, previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family. The site for this protocol is the Clinical Trials Unit in the Bristol Dental School and Hospital. Employees of the Bristol Dental School and Hospital not associated with the Clinical Trials Unit are eligible to participate
* Any participant who, in the judgement of the investigator, should not participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bristol, United Kingdom

REFERENCES:
- [Derived] West NX, Seong J, Hellin N, Macdonald EL, Jones SB, Creeth JE. Assessment of tubule occlusion properties of an experimental stannous fluoride toothpaste: A randomised clinical in situ study. J Dent. 2018 Sep;76:125-131. doi: 10.1016/j.jdent.2018.07.001. Epub 2018 Jul 5. PMID 29981778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center at United Kingdom.
Pre-assignment Details: A total of 26 participants were screened, out of which 24 participants were randomized to the study and 2 participants withdrawn their consent.
Groups:
- Test /Negative Control/Reference: Firstly, participants received dentifrice containing 0.454% stannous fluoride (test), secondly mineral water (negative control) and thirdly dentifrice containing 0.76% sodium monofluorophosphate (reference). Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 milliliters (mL) of mineral water for 5 seconds.
- Test/Reference/Negative Control: Firstly, participants received test dentifrice, secondly reference dentifrice and thirdly negative control. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Negative Control/Test/Reference: Firstly, participants received negative control, secondly test dentifrice and thirdly reference dentifrice. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Negative Control/Reference/Test: Firstly, participants received negative control, secondly reference dentifrice and thirdly test dentifrice. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Reference/Test/Negative Control: Firstly, participants received reference dentifrice, secondly test dentifrice and thirdly negative control. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Reference/Negative Control/Test: Firstly, participants received reference dentifrice, secondly negative control and thirdly test dentrifrice. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
Period: Period 1
Arm/Group | Test /Negative Control/Reference | Test/Reference/Negative Control | Negative Control/Test/Reference | Negative Control/Reference/Test | Reference/Test/Negative Control | Reference/Negative Control/Test
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Test /Negative Control/Reference | Test/Reference/Negative Control | Negative Control/Test/Reference | Negative Control/Reference/Test | Reference/Test/Negative Control | Reference/Negative Control/Test
Started | 4 | 4 | 4 | 3 | 4 | 4
Completed | 3 | 4 | 4 | 3 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other (Reason not specified) | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Test /Negative Control/Reference | Test/Reference/Negative Control | Negative Control/Test/Reference | Negative Control/Reference/Test | Reference/Test/Negative Control | Reference/Negative Control/Test
Started | 3 | 4 | 4 | 3 | 4 | 4
Completed | 3 | 3 | 4 | 3 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other (Reason not specified) | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included for baseline evaluation
Groups:
- All Randomized Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Occlusion Scores After 8 Days Treatment Application
Description: Change from baseline (pre-dose) in the mean occlusion classification score was calculated. The degree of occlusion was measured using the following classification grades; 0 Not Evaluable, 1 Occluded, 2 Mostly Occluded, 3 Equally Occluded/Unoccluded, 4 Mostly Unoccluded and 5 Unoccluded
Time Frame: Baseline and Day 8
Population: Per protocol (PP) Population was the primary analysis population, defined as those participants in the ITT (Intent to treat) population for whom all post baseline scanning electron microscopy (SEM) image scores were not deemed to be affected by protocol violations.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test Product: Participants used dentifrice containing 0.454% stannous fluoride. Appliances were brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Reference Product: Participants used dentifrice containing 0.76% sodium monofluorophosphate. Appliances brushed ex situ in 1:3 slurry of freshly prepared dentifrice twice daily then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in a 1:3 slurry of assigned dentifrice. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
- Negative Control: Participants used commercially available mineral water. Appliances brushed ex situ in mineral water twice daily were then returned to the participant's mouth. Each appliance was brushed for 1 minute (2 minutes total for both of the participant's appliances) using an electric toothbrush in mineral water. Appliances were returned to the participant's mouth and the participants rinsed with 10 mL of mineral water for 5 seconds.
Arm/Group | Test Product | Reference Product | Negative Control
Number analyzed (Participants) | 23 | 22 | 24
Score on a scale
  Pre-dose (Baseline) | 4.38 (0.383) | 4.32 (0.518) | 4.36 (0.398)
  Post-dose (Post Baseline) | 3.43 (0.760) | 3.42 (0.754) | 3.53 (0.865)
  Change | -0.95 (0.925) | -0.90 (0.933) | -0.83 (0.849)
Statistical Analysis 1: Comparison: Test Product vs Negative Control; Test type: Superiority; p = 0.5512, Mixed Models Analysis — From the MMRM model with change from pre-dose as response, participant as a random effect; and treatment, period, day, location of sample in mouth (left or right) and treatment×day interaction as fixed effects; pre-dose mean SEM score as covariate; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.46 to 0.25] — Difference is the first named treatment minus second named treatment such that a negative difference favours the first named treatment
Statistical Analysis 2: Comparison: Test Product vs Reference Product; Test type: Superiority; p = 0.9671, Mixed Models Analysis — From the MMRM model with change from pre-dose as response, subject as a random effect; and treatment, period, day, location of sample in mouth (left or right) and treatment×day interaction as fixed effects; pre-dose mean SEM score as covariate; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.36 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Reference Product vs Negative Control; Test type: Superiority; p = 0.5830, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.46 to 0.26] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Mean Occlusion Scores After 1, 4, & 10 Days Treatment Application
Description: as for outcome 1
Time Frame: Baseline, Day 1, 4, and 10
Population: PP Population was the primary analysis population, defined as those participants in the ITT (Intent to treat) population for whom all post baseline scanning electron microscopy (SEM) image scores were not deemed to be affected by protocol violations.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product | Reference Product | Negative Control
Number analyzed (Participants) | 23 | 22 | 24
Score on a scale
  Day 1: Pre-dose (Baseline) | 4.30 (0.424) | 4.38 (0.364) | 4.30 (0.486)
  Day 1: Post-dose (Post Baseline) | 3.96 (0.578) | 4.13 (0.769) | 3.86 (0.961)
  Day 1: Change from Baseline | -0.34 (0.723) | -0.26 (0.748) | -0.44 (0.876)
  Day 4: Pre-dose (Baseline) | 4.41 (0.465) | 4.30 (0.466) | 4.23 (0.404)
  Day 4: Post-dose (Post Baseline) | 3.51 (0.825) | 3.60 (0.843) | 3.98 (0.762)
  Day 4: Change from Baseline | -0.91 (0.819) | -0.70 (0.875) | -0.25 (0.827)
  Day 10: Pre-dose (Baseline) | 4.31 (0.410) | 4.31 (0.418) | 4.36 (0.428)
  Day 10: Post-dose (Post Baseline) | 3.13 (0.958) | 3.49 (0.841) | 3.74 (0.862)
  Day 10: Change from Baseline | -1.18 (0.910) | -0.82 (0.827) | -0.62 (0.958)

ADVERSE EVENTS:
Time Frame: Baseline to Day 10
Arm/Group | Test Product | Reference Product | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 2/23 | 4/22 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=23) | Reference Product (N=22) | Negative Control (N=24)
Sensitivity of Teeth (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 0 | 1 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 2
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.